CLINICAL TRIAL: NCT03377062
Title: Cerebrovascular Accident (CVA) in Patients Suffering From Decreased Consciousness, Confusion or Headaches to an Emergency Room
Brief Title: CVA in Patients Suffering From Decreased Consciousness, Confusion or Headaches to an Emergency Room
Status: Not yet recruiting | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dana Baron Shahaf, MD PhD, Primary Investigator, Rambam Health Care Campus
Other Study IDs: 260-16
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: CVA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EEG monitoring: Patients arriving to the emergency room with decreased consciousness, severe headaches or dizziness
  Interventions: Diagnostic Test: EEG monitoring

INTERVENTIONS:
Diagnostic Test: EEG monitoring — Five-minute of EEG monitoring accompanied with auditory stimulation.

SUMMARY:
A CVA occurs when there is a sudden interruption of blood supply to the brain. Fast identification of CVA is crucial in order to refer the patient to an appropriate medical center as well as to direct him/her to a suitable treatment upon arrival to the Medical Center, in order to minimize the permanent damage to the brain. In this study, we are evaluating a tool for detecting CVA based on EEG (electroencephalograph) data analysis using innovative algorithm. The system is comprised of four electrodes, reference electrode and earphones for auditory stimulation. In the study, 120 patients arriving to the emergency room with decreased consciousness, severe headaches or dizziness will be monitored for five-minute each, with EEG accompanied with auditory stimulation. The EEG analysis will be performed based on the synchronization of the front and back hemispheres. During CVA, specific hemisphere is damaged, therefore desynchronization is expected. The purpose of this study is to develop a tool for identifying CVA in patients who have no clear CVA related signs.

ELIGIBILITY:
Inclusion Criteria:

Patients arriving to the emergency room with decreased consciousness, severe headaches or dizziness

Exclusion Criteria:

Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients arriving to the emergency room with decreased consciousness, severe headaches or dizziness
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Desynchronization Index | 1 day
  Desynchronization Index calculated from EEG data correlation with CVA events

SECONDARY OUTCOMES:
EEG variablity | 1 day
  EEG variability will be evaluated in correlation to various medical measures (ECG, hypoglycemic state, hypothermia)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel